CLINICAL TRIAL: NCT00809289
Title: A Randomized, Multiple Dose, Placebo and Active Controlled 3-way Crossover Study to Investigate the Effects of Esreboxetine on QTc Interval in Healthy Volunteers
Brief Title: Phase 1 Thorough QT (TQT) Study in Young Healthy Volunteers
Acronym: TQT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A6061065
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Fibromyalgia
Keywords: Thorough QT/QTc study
MeSH Terms: conditions — Fibromyalgia | interventions — esreboxetine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- One (Experimental)
  Interventions: Drug: esreboxetine
- Two (Placebo Comparator)
  Interventions: Drug: placebo
- Three (Active Comparator): Administration of a single oral dse of 400mg moxifloxacin
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: esreboxetine — Once daily administration of 4mg esreboxetine for 3 days, followed by 8mg esreboxetine for 3 days, followed by 10mg esreboxetine for 3 days. Drug will be administered double-blind.
  Arms: One
Drug: placebo — Once daily administration of placebo for 9 days. Placebo will be administered double blind
  Arms: Two
Drug: moxifloxacin — Once daily administration of placebo for 8 days followed by open label single oral dose of 400mg moxifloxacin on day 9
  Arms: Three

SUMMARY:
This Phase 1 study will assess the effects of esreboxetine on the heart. In particular the effects on a specific electrocardiogram (ECG) measurement called QTc will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 55 years
* Body mass Index of approximately 18 to 30kg/m2
* Informed consent document signed by the subject or a legally acceptable representative
* Subjects who are willing and able to comply with the scheduled visits, treatment tests, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic psychiatric, neurologic or allergic disease or clinical findings at screening
* Conditions possibly affecting drug absorption
* 12-lead ECg demonstrating QTc > 450ms or any other clinically significant abnormalities at screen
* Positive urine drug screen
* Hypersensitivity to moxifloxacin
* Unwilling or unable to comply with the lifestyle guidelines in the protocol Treatment with an investigational drug within 3 months or 5 half lives (whichever is longer) preceding the first dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To assess whether multiple dose administration of esreboxetine has the potential to affect QTc in healthy volunteers | Up to 24 hours

SECONDARY OUTCOMES:
To asses the the relationship between plasma concentrations of esreboxetine and its effects, if any on the QTc interval | Up to 24 hours
To assess the effects of a positive control (moxifloxacin) on QTc interval in healthy volunteers | Up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061065&StudyName=Phase%201%20thorough%20QT%20%28TQT%29%20study%20in%20young%20healthy%20volunteers